CLINICAL TRIAL: NCT06542393
Title: Patient Blood Manegement (PBM) as Perioperative Strategy to Anemic Patients Who Will be Submitted to Coronary Artery Bypass Graft (CABG).
Brief Title: PBM as Strategy to CABG Anemic Patients Bypass Graft (CABG)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, LEONARDO OHASHI, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0009/2023
Record Dates: First submitted 2024-07-09; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Anemia; Coronary Disease; Coronary Artery Disease; Coronary Stenosis; Coronary Occlusion; Systemic Inflammatory Response; Bleeding; Epigenetic Disorder
MeSH Terms: conditions — Anemia; Coronary Disease; Coronary Artery Disease; Coronary Stenosis; Coronary Occlusion; Hemorrhage | interventions — Erythropoietin; Blood Transfusion

STUDY DESIGN:
Intervention Model Description: Randomized (intervention group) for anemic patients Non-randomized (control group) for non-anemic patients
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized Anemia Group for non-PBM protocol (GNPBM) (Experimental): Patients > 18 years admitted to Hospital São Paulo for Coronary Artery Bypass Grafting (CABG) surgery who are hospitalized in the Cardiovascular Surgery department or another specialty unit and are anemic (Hemoglobin - Hb < 12g/dl in women and < 13g/dl in men)
  Interventions: Procedure: blood transfusion
- Randomized Anemia Group for PBM protocol (GPBM) (Experimental): Patients >18 years admitted to Hospital São Paulo for Coronary Artery Bypass Grafting (CABG) surgery who are hospitalized in the Cardiovascular Surgery department or another specialty unit and are anemic (Hb < 12g/dl in women and < 13g/dl in men)
  Interventions: Drug: Erythropoietin
- Control Group (GC) (No Intervention): Patients > 18 years admitted to Hospital SãoPaulo for Coronary Artery Bypass Grafting (CABG) surgery who arehospitalized in the Cardiovascular Surgery department or another specialty unit and do not have anemia (Hb > 13g/dl in men and > 12g/dl in women)

INTERVENTIONS:
Drug: Erythropoietin — * Treatment regimen for hospitalized patients awaiting non-urgent surgeries: Administer EPO 600 IU/kg/week via subcutaneous (SC) or intravenous (IV) route, followed by 300 IU/kg/day via SC or IV 10 days before surgery. If ferritin < 100 ng/dL, supplement with IV iron (Iron hydroxide up to 600 mg/week or Ferric carboxymaltose up to 1000 mg/week).
  * Treatment regimen for hospitalized patients awaiting non-urgent surgeries with less than 5 days until surgery: Administer 40000 UI of EPO intravenous (IV) attack and supplement with IV iron (Iron hydroxide up to 600 mg/week or Ferric carboxymaltose up to 2000 mg/week), then 300UI/Kg/day IV or SC of EPO until day of surgery.
  Arms: Randomized Anemia Group for PBM protocol (GPBM)
Procedure: blood transfusion — After surgery, this group will receive one unit of RBC at the moment of ICU admission.
  Hb > 8 g/dl: 1 unit of RBC. HB < 8 g/dl: 2 units of RBC.
  Arms: Randomized Anemia Group for non-PBM protocol (GNPBM)

SUMMARY:
Anemia poses risks during coronary artery bypass grafting (CABG), increasing complications and mortality rates. Blood transfusions in cardiac surgery have negative outcomes, prompting the use of erythropoietin in Patient Blood Management (PBM) to limit transfusion needs and enhance postoperative recovery. EPO can reduce blood component requirements, adverse events, and inflammation in anemic CABG patients. A study aims to minimize transfusions through a PBM anemia treatment protocol for CABG patients, comparing outcomes in three groups: a Control Group (CG), a Non-PBM Group (NPBMG) treated with blood components, and a PBM Group (GPBM) treated with EPO. Parameters include post-op stay, mortality, cardiovascular events, non-cardiovascular events, ICU time, mechanical ventilation duration, vasoactive drug use, inflammatory responses, and cardiac cell death. Analysis will consider demographic and clinical factors, with expectations that GPBM will yield superior results compared to NPBMG and similar or better outcomes than CG.

DETAILED DESCRIPTION:
Anemia increases the risk of postoperative complications and mortality in patients undergoing coronary artery bypass grafting (CABG). In addition, the use of blood transfusions during cardiac surgery is associated with adverse effects and unfavorable outcomes. To reduce the need for transfusions and improve post-operative results, erythropoietin is used as part of Patient Blood Management (PBM). In anemic patients undergoing CABG, the use of Erythropoietin (EPO) can eliminate the need for blood components during and after surgery, as well as reduce adverse events and inflammation. The objectives of the proposed study are to reduce or eliminate the number of transfusions in the intraoperative and postoperative context by means of a Patient Blood Management (PBM) anemia treatment protocol for anemic patients who will undergo Coronary Artery Bypass Graft Surgery (CABG). The proposed study is a prospective, non-controlled interventional study to be carried out with anemic patients awaiting CABG surgery at Hospital São Paulo. There will be three groups of 40 participants each: Control Group (CG) of non-anemic individuals preoperatively; Non- PBM Group (NPBMG) of anemic individuals preoperatively and treated with blood components according to need; PBM Group (GPBM) of anemic individuals preoperatively and treated with EPO. The following parameters will be compared: length of postoperative hospital stay; mortality; postoperative cardiovascular events: clinical stroke, perioperative infarction, surgical reoperation due to bleeding; non- cardiovascular events: surgical site-associated infection and acute renal dysfunction; time in postoperative intensive care; time on mechanical ventilation; need for vasoactive drug use; inflammatory process and intra- and postoperative cardiac cell death. Confounding factors such as demographic and clinical parameters will be included in the analysis. It is expected that the GPBM will obtain the best results in relation to the GNPBM, similar to or better than the CG.

ELIGIBILITY:
Inclusion Criteria:

* Eletive surgery;
* Only CABG as procedure;
* Off pump CABG candidate.

Exclusion Criteria:

* Age > 80 years;
* Chronic dialytic kidney disease;
* Chronic rheumatologic disease;
* Men with Hb levels > 13 g/dl and < 8g/dl;
* Women with Hb levels > 12 g/dl and < 8g/dl;
* Presence of another heart disease requiring surgical intervention;
* Presence of hepatic insufficiency;
* Presence of any implantable electronic cardiac device in any cardiac chambers;
* Pregnancy;
* Diagnosis of malignant neoplasia;
* Thrombophilias;
* Need for Erythropoietin treatment due to any other disease.
* Recent ischemic event (< 3 months).
* Ejection fraction <30%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of units of Red Blood Cells (RBC) | Until perioperative day 3
  Compare the need of blood transfusion in the perioperative period

SECONDARY OUTCOMES:
Length of ICU stay | From time of admission after surgery to time of clinical conditions of discharge (time of ICU medical discharge, not time of ICU room exit). Up to 240 hours.
  Hours
Length of hospital stay | From time of ICU medical discharge until time of Hospital discharge (Up to 14 days).
  Days
Length of mechanical ventilation | From time of intubation by anesthesia team until time of extubation by ICU team (Up to 240 hours).
  Hours
Need of Dyalisis (Acute Kidney Disease) | Based on KDIGO classification of Acute Kdney Injury, level III of the classification. (Up to 120 hours from ICU admission, accountable from the time Dyalisis is indicated).
  Needing of dyalisis in peoperative period
Perioperative infection | Until perioperative day 3
  Anytype
Bleeding | From time of admission on ICU until hour 24th after admission (accountable amount from how many chest tubes the patient was admitted).
  Thorax drain tubes bleeding (ml)
Epigenetics alterations | Until perioperative day 3
  . Differentially methylated regions (DMRs) and differentially methylated loci (DMLs) will be considered to determine if these regions are hypermethylated or hypomethylated in the comparison between groups.
Inflammatory response | Until perioperative day 3
  A total of 25 μl of serum per patient will be used for the detection of the following analytes: IL-1β, IL-6, IL-10, TNF-α, CRP, and NT-ProBNP.
Perioperative myocardial infarction | Until perioperative day 3
  According to type 5 Myocardial ischemia
Stroke | Until perioperative day 3
  Any level of neurological deficit
Hemoglobin levels | Until perioperative day 3 and at discharge
  Accountable in g/dl
All-cause mortality | From day of the intervention (if intervention group) or from the moment of surgery (if control group) until day of hospital discharge (death from any cause accountable as in-hospital mortality).
  Death from any cause accountable as in-hospital mortality
Cardiovascular mortality | From day of the intervention (if intervention group) or from the moment of surgery (if control group) until day of hospital discharge (any cardiovascular reason as main cause of death accountable as in-hospital mortality).)
  any cardiovascular reason as main cause of death accountable as in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Leonardo Ohashi, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghamdi AA, Albanna MJ, Guru V, Brister SJ. Does the use of erythropoietin reduce the risk of exposure to allogeneic blood transfusion in cardiac surgery? A systematic review and meta-analysis. J Card Surg. 2006 May-Jun;21(3):320-6. doi: 10.1111/j.1540-8191.2006.00241.x. PMID 16684074
- [Background] Althoff FC, Neb H, Herrmann E, Trentino KM, Vernich L, Fullenbach C, Freedman J, Waters JH, Farmer S, Leahy MF, Zacharowski K, Meybohm P, Choorapoikayil S. Multimodal Patient Blood Management Program Based on a Three-pillar Strategy: A Systematic Review and Meta-analysis. Ann Surg. 2019 May;269(5):794-804. doi: 10.1097/SLA.0000000000003095. PMID 30418206
- [Background] Anthes E. Evidence-based medicine: Save blood, save lives. Nature. 2015 Apr 2;520(7545):24-6. doi: 10.1038/520024a. No abstract available. PMID 25832389
- [Background] Bian XX, Yuan XS, Qi CP. Effect of recombinant human erythropoietin on serum S100B protein and interleukin-6 levels after traumatic brain injury in the rat. Neurol Med Chir (Tokyo). 2010;50(5):361-6. doi: 10.2176/nmc.50.361. PMID 20505289
- [Background] Avni T, Bieber A, Grossman A, Green H, Leibovici L, Gafter-Gvili A. The safety of intravenous iron preparations: systematic review and meta-analysis. Mayo Clin Proc. 2015 Jan;90(1):12-23. doi: 10.1016/j.mayocp.2014.10.007. Epub 2014 Oct 30. PMID 25572192
- [Background] Bogoyevitch MA. An update on the cardiac effects of erythropoietin cardioprotection by erythropoietin and the lessons learnt from studies in neuroprotection. Cardiovasc Res. 2004 Aug 1;63(2):208-16. doi: 10.1016/j.cardiores.2004.03.017. PMID 15249178
- [Background] Cho BC, Serini J, Zorrilla-Vaca A, Scott MJ, Gehrie EA, Frank SM, Grant MC. Impact of Preoperative Erythropoietin on Allogeneic Blood Transfusions in Surgical Patients: Results From a Systematic Review and Meta-analysis. Anesth Analg. 2019 May;128(5):981-992. doi: 10.1213/ANE.0000000000004005. PMID 30649068
- [Background] Engoren MC, Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ. Effect of blood transfusion on long-term survival after cardiac operation. Ann Thorac Surg. 2002 Oct;74(4):1180-6. doi: 10.1016/s0003-4975(02)03766-9. PMID 12400765
- [Background] Farmer SL, Towler SC, Leahy MF, Hofmann A. Drivers for change: Western Australia Patient Blood Management Program (WA PBMP), World Health Assembly (WHA) and Advisory Committee on Blood Safety and Availability (ACBSA). Best Pract Res Clin Anaesthesiol. 2013 Mar;27(1):43-58. doi: 10.1016/j.bpa.2012.12.007. PMID 23590915
- [Background] Ferrario M, Arbustini E, Massa M, Rosti V, Marziliano N, Raineri C, Campanelli R, Bertoletti A, De Ferrari GM, Klersy C, Angoli L, Bramucci E, Marinoni B, Ferlini M, Moretti E, Raisaro A, Repetto A, Schwartz PJ, Tavazzi L. High-dose erythropoietin in patients with acute myocardial infarction: a pilot, randomised, placebo-controlled study. Int J Cardiol. 2011 Feb 17;147(1):124-31. doi: 10.1016/j.ijcard.2009.10.028. Epub 2009 Nov 10. PMID 19906454
- [Background] Haljan G, Maitland A, Buchan A, Arora RC, King M, Haigh J, Culleton B, Faris P, Zygun D. The erythropoietin neuroprotective effect: assessment in CABG surgery (TENPEAKS): a randomized, double-blind, placebo controlled, proof-of-concept clinical trial. Stroke. 2009 Aug;40(8):2769-75. doi: 10.1161/STROKEAHA.109.549436. Epub 2009 Jun 25. PMID 19556536
- [Background] Hayden SJ, Albert TJ, Watkins TR, Swenson ER. Anemia in critical illness: insights into etiology, consequences, and management. Am J Respir Crit Care Med. 2012 May 15;185(10):1049-57. doi: 10.1164/rccm.201110-1915CI. Epub 2012 Jan 26. PMID 22281832
- [Background] Hogan M, Klein AA, Richards T. The impact of anaemia and intravenous iron replacement therapy on outcomes in cardiac surgery. Eur J Cardiothorac Surg. 2015 Feb;47(2):218-26. doi: 10.1093/ejcts/ezu200. Epub 2014 May 13. PMID 24824650
- [Background] Jadwin DF, Fenderson PG, Friedman MT, Jenkins I, Shander A, Waters JH, Friedman A, Tesoriero E, Refaai MA, Shih AW, Awan T, Ngo AL, Perez JA, Reynolds JD. Determination of Unnecessary Blood Transfusion by Comprehensive 15-Hospital Record Review. Jt Comm J Qual Patient Saf. 2023 Jan;49(1):42-52. doi: 10.1016/j.jcjq.2022.10.006. Epub 2022 Nov 8. PMID 36494267
- [Background] Lin DM, Lin ES, Tran MH. Efficacy and safety of erythropoietin and intravenous iron in perioperative blood management: a systematic review. Transfus Med Rev. 2013 Oct;27(4):221-34. doi: 10.1016/j.tmrv.2013.09.001. Epub 2013 Oct 15. PMID 24135037
- [Background] Lipsic E, van der Meer P, Voors AA, Westenbrink BD, van den Heuvel AF, de Boer HC, van Zonneveld AJ, Schoemaker RG, van Gilst WH, Zijlstra F, van Veldhuisen DJ. A single bolus of a long-acting erythropoietin analogue darbepoetin alfa in patients with acute myocardial infarction: a randomized feasibility and safety study. Cardiovasc Drugs Ther. 2006 Apr;20(2):135-41. doi: 10.1007/s10557-006-7680-5. PMID 16761193
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785
- [Background] Kulier A, Levin J, Moser R, Rumpold-Seitlinger G, Tudor IC, Snyder-Ramos SA, Moehnle P, Mangano DT; Investigators of the Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Impact of preoperative anemia on outcome in patients undergoing coronary artery bypass graft surgery. Circulation. 2007 Jul 31;116(5):471-9. doi: 10.1161/CIRCULATIONAHA.106.653501. Epub 2007 Jul 9. PMID 17620512
- [Background] Mathias JM. Safety, cost savings, simplicity back broader use of bloodless surgery. OR Manager. 2013 May;29(5):1, 6, 8-9. No abstract available. PMID 23755462
- [Background] Menkis AH, Martin J, Cheng DC, Fitzgerald DC, Freedman JJ, Gao C, Koster A, Mackenzie GS, Murphy GJ, Spiess B, Ad N. Drug, devices, technologies, and techniques for blood management in minimally invasive and conventional cardiothoracic surgery: a consensus statement from the International Society for Minimally Invasive Cardiothoracic Surgery (ISMICS) 2011. Innovations (Phila). 2012 Jul-Aug;7(4):229-41. doi: 10.1097/IMI.0b013e3182747699. PMID 23123988
- [Background] Murphy MF, Goodnough LT. The scientific basis for patient blood management. Transfus Clin Biol. 2015 Aug;22(3):90-6. doi: 10.1016/j.tracli.2015.04.001. Epub 2015 May 8. PMID 25959997
- [Background] Munoz M, Acheson AG, Auerbach M, Besser M, Habler O, Kehlet H, Liumbruno GM, Lasocki S, Meybohm P, Rao Baikady R, Richards T, Shander A, So-Osman C, Spahn DR, Klein AA. International consensus statement on the peri-operative management of anaemia and iron deficiency. Anaesthesia. 2017 Feb;72(2):233-247. doi: 10.1111/anae.13773. Epub 2016 Dec 20. PMID 27996086
- [Background] Neumann FJ, Sousa-Uva M. 'Ten commandments' for the 2018 ESC/EACTS Guidelines on Myocardial Revascularization. Eur Heart J. 2019 Jan 7;40(2):79-80. doi: 10.1093/eurheartj/ehy855. No abstract available. PMID 30615155
- [Background] Oh SW, Chin HJ, Chae DW, Na KY. Erythropoietin improves long-term outcomes in patients with acute kidney injury after coronary artery bypass grafting. J Korean Med Sci. 2012 May;27(5):506-11. doi: 10.3346/jkms.2012.27.5.506. Epub 2012 Apr 25. PMID 22563215
- [Background] Ozawa T, Toba K, Suzuki H, Kato K, Iso Y, Akutsu Y, Kobayashi Y, Takeyama Y, Kobayashi N, Yoshimura N, Akazawa K, Aizawa Y; EPO/AMI-I Pilot Study Researchers. Single-dose intravenous administration of recombinant human erythropoietin is a promising treatment for patients with acute myocardial infarction - randomized controlled pilot trial of EPO/AMI-1 study -. Circ J. 2010 Jul;74(7):1415-23. doi: 10.1253/circj.cj-10-0109. Epub 2010 May 22. PMID 20501957
- [Background] Paone G, Likosky DS, Brewer R, Theurer PF, Bell GF, Cogan CM, Prager RL; Membership of the Michigan Society of Thoracic and Cardiovascular Surgeons. Transfusion of 1 and 2 units of red blood cells is associated with increased morbidity and mortality. Ann Thorac Surg. 2014 Jan;97(1):87-93; discussion 93-4. doi: 10.1016/j.athoracsur.2013.07.020. Epub 2013 Oct 3. PMID 24094521
- [Background] Pavenski K, Howell A, Mazer CD, Hare GMT, Freedman J. ONTraC: A 20-Year History of a Successfully Coordinated Provincewide Patient Blood Management Program: Lessons Learned and Goals Achieved. Anesth Analg. 2022 Sep 1;135(3):448-458. doi: 10.1213/ANE.0000000000006065. Epub 2022 Aug 17. PMID 35977355
- [Background] Pieracci FM, Henderson P, Rodney JR, Holena DN, Genisca A, Ip I, Benkert S, Hydo LJ, Eachempati SR, Shou J, Barie PS. Randomized, double-blind, placebo-controlled trial of effects of enteral iron supplementation on anemia and risk of infection during surgical critical illness. Surg Infect (Larchmt). 2009 Feb;10(1):9-19. doi: 10.1089/sur.2008.043. PMID 19245362
- [Background] Poulsen TD, Andersen LW, Steinbruchel D, Gotze JP, Jorgensen OS, Olsen NV. Two large preoperative doses of erythropoietin do not reduce the systemic inflammatory response to cardiac surgery. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):316-23. doi: 10.1053/j.jvca.2008.08.018. Epub 2008 Oct 22. PMID 18948032
- [Background] Santos AA, Silva JP, Silva Lda F, Sousa AG, Piotto RF, Baumgratz JF. Therapeutic options to minimize allogeneic blood transfusions and their adverse effects in cardiac surgery: a systematic review. Rev Bras Cir Cardiovasc. 2014 Oct-Dec;29(4):606-21. doi: 10.5935/1678-9741.20140114. PMID 25714216
- [Background] Shander A, Isbister J, Gombotz H. Patient blood management: the global view. Transfusion. 2016 Mar;56 Suppl 1:S94-102. doi: 10.1111/trf.13529. No abstract available. PMID 27001367
- [Background] Suh JW, Yoon YE, Oh IY, Yoon CH, Cho YS, Youn TJ, Chae IH, Choi DJ. A single-center prospective randomized controlled trial evaluating the safety and efficacy of IntraCoronary Erythropoietin delivery BEfore Reperfusion: gauging infarct size in patients with acute ST-segment elevation myocardial infarction. Study design and rationale of the 'ICEBERG Trial'. Contemp Clin Trials. 2013 May;35(1):145-50. doi: 10.1016/j.cct.2013.03.001. Epub 2013 Mar 16. PMID 23506972
- [Background] Tan GM, Guinn NR, Frank SM, Shander A. Proceedings From the Society for Advancement of Blood Management Annual Meeting 2017: Management Dilemmas of the Surgical Patient-When Blood Is Not an Option. Anesth Analg. 2019 Jan;128(1):144-151. doi: 10.1213/ANE.0000000000003478. PMID 29958216
- [Background] Tang M, Ravn HB, Andreasen JJ, Greisen J, Thomassen S, Fabrin A, Jakobsen CJ. Fewer transfusions are still more-red blood cell transfusions affect long-term mortality in cardiac surgery. Eur J Cardiothorac Surg. 2023 Apr 3;63(4):ezad101. doi: 10.1093/ejcts/ezad101. PMID 36943381
- [Background] Taniguchi N, Nakamura T, Sawada T, Matsubara K, Furukawa K, Hadase M, Nakahara Y, Nakamura T, Matsubara H. Erythropoietin prevention trial of coronary restenosis and cardiac remodeling after ST-elevated acute myocardial infarction (EPOC-AMI): a pilot, randomized, placebo-controlled study. Circ J. 2010 Nov;74(11):2365-71. doi: 10.1253/circj.cj-10-0267. Epub 2010 Sep 8. PMID 20834185
- [Background] Tasanarong A, Duangchana S, Sumransurp S, Homvises B, Satdhabudha O. Prophylaxis with erythropoietin versus placebo reduces acute kidney injury and neutrophil gelatinase-associated lipocalin in patients undergoing cardiac surgery: a randomized, double-blind controlled trial. BMC Nephrol. 2013 Jul 5;14:136. doi: 10.1186/1471-2369-14-136. PMID 23829828
- [Background] Teringova E, Tousek P. Apoptosis in ischemic heart disease. J Transl Med. 2017 May 1;15(1):87. doi: 10.1186/s12967-017-1191-y. PMID 28460644
- [Background] Shen Y, Wang Y, Li D, Wang C, Xu B, Dong G, Huang H, Jing H. Recombinant human erythropoietin pretreatment attenuates heart ischemia-reperfusion injury in rats by suppressing the systemic inflammatory response. Transplant Proc. 2010 Jun;42(5):1595-7. doi: 10.1016/j.transproceed.2009.11.050. PMID 20620481
- [Background] Sun LJ, Qiao W, Xiao YJ, Ren WD. Layer-specific strain for assessing the effect of naringin on systolic myocardial dysfunction induced by sepsis and its underlying mechanisms. J Int Med Res. 2021 Jan;49(1):300060520986369. doi: 10.1177/0300060520986369. PMID 33445988
- [Background] Wademan BH, Galvin SD. Desmopressin for reducing postoperative blood loss and transfusion requirements following cardiac surgery in adults. Interact Cardiovasc Thorac Surg. 2014 Mar;18(3):360-70. doi: 10.1093/icvts/ivt491. Epub 2013 Nov 21. PMID 24263581
- [Background] Yang SS, Al Kharusi L, Gosselin A, Chirico A, Baradari PG, Cameron MJ. Iron supplementation for patients undergoing cardiac surgery: a systematic review and meta-analysis of randomized controlled trials. Can J Anaesth. 2022 Jan;69(1):129-139. doi: 10.1007/s12630-021-02113-z. Epub 2021 Sep 24. PMID 34559371
- [Background] Ziabakhsh-Tabary S, Jalalian R, Mokhtari-Esbuie F, Habibi MR. Echocardiographic Evaluation of the Effects of a Single Bolus of Erythropoietin on Reducing Ischemia-Reperfusion Injuries during Coronary Artery Bypass Graft Surgery; A Randomized, Double-Blind, Placebo-Control Study. Iran J Med Sci. 2014 Mar;39(2):94-101. PMID 24644377